CLINICAL TRIAL: NCT07284251
Title: A Comparison of the D Blade and Mac Blade C-MAC Video Laryngoscope for Double-Lumen Endotracheal Intubation in Patients With Predicted Normal Airways
Brief Title: C-MAC Video Laryngoscope for Double-Lumen Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, FERAY AKGUL ERDIL, Clinical Professor Doctor, Inonu University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: INU-AR-FAE-01
Record Dates: First submitted 2025-12-01; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Device Performance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group D blade (Active Comparator): DLT (with the stylet in place) was molded along the blade convexity, and sequential rotation was performed for insertion. After the bronchial lumen tip engaged the glottis, the stylet was removed, and the DLT was rotated 180° counterclockwise to facilitate passage of the bronchial cuff. The DLT was then rotated 90° clockwise to ensure it entered the left main bronchus
  Interventions: Device: C-MAC Macintosh blade Video Laryngoscope; Device: DİRECT Laryngoscopy
- Group M (Active Comparator): once the bronchial cuff had passed through the vocal cords, the double-lumen tube was inserted using the conventional method
  Interventions: Device: DİRECT Laryngoscopy; Device: D blade CMac videolaryngoscopy
- Group DL (Direct laryngoscopy macintosch blade, conventional . placebo) (Placebo Comparator): once the bronchial cuff had passed through the vocal cords, the double-lumen tube was inserted using the conventional method
  Interventions: Device: C-MAC Macintosh blade Video Laryngoscope; Device: D blade CMac videolaryngoscopy

INTERVENTIONS:
Device: C-MAC Macintosh blade Video Laryngoscope — videolaryngoscopes have been increasingly used in thoracic surgery, particularly in patients with difficult airways, as they enhance visualization of laryngeal structures and facilitate lung separationThe D-blade and Mac blade are adapted for use with the C-MAC system.10 The C-MAC Mac and D-blade may be a viable alternative to direct laryngoscopy with the Mac blade in routine practice.
  Arms: Group D blade; Group DL (Direct laryngoscopy macintosch blade, conventional . placebo)
Device: DİRECT Laryngoscopy — In patients without predicted difficult airways undergoing thoracic surgery, direct laryngoscopy with a Mac blade remains the recommended technique for DLT placement
  Arms: Group D blade; Group M
Device: D blade CMac videolaryngoscopy — videolaryngoscopes have been increasingly used in thoracic surgery, particularly in patients with difficult airways, as they enhance visualization of laryngeal structures and facilitate lung separation
  Arms: Group DL (Direct laryngoscopy macintosch blade, conventional . placebo); Group M

SUMMARY:
. The study aimed to compare the C-MAC D-Blade (Group D) and the C-MAC Macintosh blade (Group M) with the conventional direct laryngoscopy macintosh blade (Group DL) in patients with predicted normal airways undergoing thoracic surgery requiring double lumen tube (DLT) placement.

DETAILED DESCRIPTION:
The double-lumen tracheal tube (DLT) is the standard device for achieving one-lung ventilation in thoracic surgery. Compared to a single-lumen endotracheal tube, the DLT is longer, stiffer, and has a larger external diameter, making its insertion more challenging. Recently, videolaryngoscopes have been increasingly used in thoracic surgery, particularly in patients with difficult airways, as they enhance visualization of laryngeal structures and facilitate lung separation.However, the role of the videolaryngoscope in DLT intubation remains unclear due to the larger size of the DLT and the discrepancy between the curves of the DLT and the videolaryngoscope blade, which can affect vocal cord visualization and, consequently, intubation success.

Videolaryngoscopes can be classified as standard or hyperangulated based on blade angulation. The results of clinical studies on hyperangulated videolaryngoscopes for DLT placement have been inconsistent, particularly regarding intubation time. While some hyperangulated videolaryngoscopes have demonstrated superiority over the macintosh (Mac) blade laryngoscope in normal airway patients, others have not. These discrepancies may stem from the use of manikins in some studies, variations in clinician experience with videolaryngoscopes, or differences in intubation techniques.

In patients without predicted difficult airways undergoing thoracic surgery, direct laryngoscopy with a Mac blade remains the recommended technique for DLT placement. The C-MAC videolaryngoscope is designed based on the Mac blade and has been associated with improved laryngeal visualization and reduced need for additional maneuvers to facilitate intubation. The D-blade and Mac blade are adapted for use with the C-MAC system. The C-MAC Mac and D-blade may be a viable alternative to direct laryngoscopy with the Mac blade in routine practice.

This randomized controlled study aimed to compare the C-MAC D-Blade and the C-MAC Mac blade with the conventional direct laryngoscopy Mac blade in patients with predicted normal airways undergoing thoracic surgery requiring DLT placement. The primary outcome measure was intubation time. Additional parameters assessed included exposure time, the ease of intubation, number of laryngoscopy attempts, and maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) I to III,
* Patients requiring one-lung ventilation via DLT intubation

Exclusion Criteria:

* Patients with a history of difficult endotracheal intubation or mask ventilation,
* Patients with severe pulmonary ventilation dysfunction,
* Patients with a risk of pulmonary aspiration patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
intubation time | up to 10 minutes after intubation from recording
  DLT insertion time was defined as the period from when the intubation device passed the patient's lips until three complete end-tidal carbon dioxide cycles were displayed on the monitor

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz tunc ozer, doctor, Principal Investigator — Inonu University
Locations (1):
- inonu University, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No